CLINICAL TRIAL: NCT05925387
Title: The Impact of an Educational Program on Child Abuse and Neglect Knowledge and Awareness Levels Among Nursing Students: A Randomized Controlled Study
Brief Title: Educational Program's Impact on Nursing Students' Knowledge and Awareness of Child Abuse and Neglect
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: YeditepeUniversity
Record Dates: First submitted 2023-06-20; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Child Abuse; Child Neglect
Keywords: Child Abuse and Neglect; Child Maltreatment; Nursing Students' Knowledge; Nursing Students' Awareness

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Study
Who Masked: Outcomes Assessor
Masking Description: The statistician who performed the data analysis saw the experimental and control groups as group A and group B, without knowing which group was the experimental or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): All volunteers completed a pre-test, which includes an additional two scales along with the sociodemographic data form, and two post-tests, which only include the scales. Both groups will receive the Child Abuse and Neglect Awareness Training, which will last approximately 60 minutes. Both groups will complete the pre-test and post-tests at the same time. However, immediately after the pre-test, the experimental group will receive the training and then complete the 1st post-test, followed by the 2nd post-test one month later. Additionally, the second post-test will be administered to both groups simultaneously one month after the completion of the first post-test. After the completion of all the tests, the control group also received the same training, and both groups received participation certificates. Apart from these tasks, there are no other responsibilities.
  Interventions: Other: CANAP Education
- Control Group (No Intervention): Participants in the control group do not receive the intervention. They took both pretest and post-tests. The control group, on the other hand, did not receive the training but completed the first post-test simultaneously with both groups, without distinguishing between the experimental and control groups.
  They only complete online surveys. However, to follow the ethical rules, at the end of the trial, all nursing students will take the same education as their peers.

INTERVENTIONS:
Other: CANAP Education — The volunteer group included in the research consists of Yeditepe University Nursing Students. All nursing students over the age of 18, at all levels of the nursing program, will be included in the study based on voluntary participation, in accordance with the sample size. The purpose and design of the research will be explained to the 1st, 2nd, 3rd, and 4th-year nursing students. The announcement of the study will be made through Yeditepe University Nursing's social media accounts, and a consent link provided. Participants who sign the document in the consent link and upload it to the shared Google Drive received the pre-test link. Participants who complete all the procedures are provided with a participant certificate prepared by the researchers as an incentive.
  Arms: Experimental Group

SUMMARY:
Detecting and determining child abuse and neglect can be quite challenging and largely depends on the knowledge and skills of healthcare professionals. In a hospital setting, healthcare professionals frequently come across children who have experienced abuse and/or neglect. Nurses are often the first to encounter the child and their family, initiating the process of taking a medical history and establishing closer interactions during care and treatment. To accurately recognize the case and provide appropriate care using the right approach, nurses need to possess sufficient knowledge and skills related to child abuse and neglect. The lack of adequate education on child abuse and neglect, as well as insufficient research on the subject, can lead to a lack of information and cases being overlooked. To identify and report cases of child abuse and neglect, it is important for nurses, especially before starting their profession, to have a sufficient level of knowledge about the signs and risks of child abuse and neglect. This study aims to examine the impact of an educational program targeting nursing students on their knowledge and awareness levels regarding child abuse and neglect.

DETAILED DESCRIPTION:
Detecting and identifying child abuse and neglect is quite challenging and relies heavily on the knowledge and skills of healthcare professionals (Child Welfare Information Gateway, 2019). In a hospital setting, healthcare professionals frequently encounter children who have experienced abuse and/or neglect. Nurses, who are often the first to interact with the child and their family, play a crucial role starting from the process of taking the medical history to provide care and treatment (Chen et al., 2022). Nurses who have frequent contact with children and their families are in a good position to protect children from abuse and neglect (Bahrami et al., 2021). Particularly in emergency departments, nurses often come across child abuse and neglect, including various types such as Munchausen by Proxy Syndrome, which is a form of physical abuse (Chen et al., 2022). Therefore, it is crucial, especially for nurses, to carefully observe children who may be victims of abuse and evaluate all children who come to the hospital for signs of abuse and neglect (Başdaş & Bozdağ, 2018). Nurses need to have sufficient knowledge and skills regarding child abuse and neglect to accurately identify cases and provide appropriate care (Jordan & Moore-Nadler, 2014). They should establish communication with the child and their family, attempt to recognize the signs and symptoms of abuse and neglect, and report the case from a forensic perspective (Chen et al., 2022). To fulfill these roles and responsibilities adequately, nurses need to receive education on child abuse and neglect (Topçu et al., 2022). Insufficient education on child abuse and neglect, as well as inadequate research on the subject, can lead to a lack of knowledge and cases being overlooked. For example, in Turkey, there are only a limited number of universities offering elective courses on child abuse and neglect within nursing curricula (Topçu et al., 2022). Similarly, a limited number of studies have shown that the level of awareness regarding child abuse and neglect is good when it is included in the pediatric nursing curriculum (Özçevik et al., 2018). However, studies conducted in Turkey involving nurses (Başdaş & Bozdağ, 2018; Burç & Güdücü Tüfekci, 2015) and particularly nursing students (Erkut et al., 2021; Ozbey et al., 2018; Seferoğlu et al., 2019; Tek & Karataş, 2021) have revealed that their knowledge levels regarding child abuse and neglect are insufficient, similar to countries like India (Poreddi et al., 2016). In order to identify cases of child abuse and neglect, it is essential for nurses, especially before entering the profession, to have sufficient knowledge about the signs and risks of child abuse and neglect. It has been emphasized that nursing students need to learn their legal responsibilities and receive education to enhance their knowledge and become more competent (Akcan & Demiralay, 2016; Bağ & Bozkurt, 2021; Kuşlu & Bulut, 2021; Seferoğlu et al., 2019).

ELIGIBILITY:
Inclusion Criteria:

* 1st, 2nd, 3rd, and 4th Grade Undergraduate Nursing Students between the ages of 18-30.
* Being a volunteer,
* Not having any disability,
* Being Turkish literate,
* Having Internet access and a Google account,
* Signing the informed consent form

Exclusion Criteria:

* Being outside the age range,
* Being a prep class student, being illiterate in Turkish

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Child Abuse and Neglect Awareness Scale (CANA-S) | Pretest
  CANA-S has 4 sub-dimensions: physical abuse, sexual abuse, emotional abuse and neglect. It consists of 20 items in total, 11 of which are reverse scored (1,2,3,5,7,10,12,13,16,17,18). It is a 5-point Likert-type scale (ranging from 1 to 5 (between "strongly disagree" and "strongly agree"). The highest score to be obtained from the scale is 100 and the lowest score is 20. Each of the subscales is 25 points. As the scores obtained from the scale increase, the level of awareness of child abuse and neglect increases; As the scores decrease, the level of awareness of child abuse and neglect decreases. In the internal consistency analysis for reliability, the Cronbach alpha value of CANA-S was found to be 0.768.
Child Abuse and Neglect Awareness Scale (CANA-S) | Immediately after the intervention
  CANA-S has 4 sub-dimensions: physical abuse, sexual abuse, emotional abuse and neglect. It consists of 20 items in total, 11 of which are reverse scored (1,2,3,5,7,10,12,13,16,17,18). It is a 5-point Likert-type scale (ranging from 1 to 5 (between "strongly disagree" and "strongly agree"). The highest score to be obtained from the scale is 100 and the lowest score is 20. Each of the subscales is 25 points. As the scores obtained from the scale increase, the level of awareness of child abuse and neglect increases; As the scores decrease, the level of awareness of child abuse and neglect decreases. In the internal consistency analysis for reliability, the Cronbach alpha value of CANA-S was found to be 0.768.
Child Abuse and Neglect Awareness Scale (CANA-S) | 1 month after the intervention
  CANA-S has 4 sub-dimensions: physical abuse, sexual abuse, emotional abuse and neglect. It consists of 20 items in total, 11 of which are reverse scored (1,2,3,5,7,10,12,13,16,17,18). It is a 5-point Likert-type scale (ranging from 1 to 5 (between "strongly disagree" and "strongly agree"). The highest score to be obtained from the scale is 100 and the lowest score is 20. Each of the subscales is 25 points. As the scores obtained from the scale increase, the level of awareness of child abuse and neglect increases; As the scores decrease, the level of awareness of child abuse and neglect decreases. In the internal consistency analysis for reliability, the Cronbach alpha value of CANA-S was found to be 0.768.

SECONDARY OUTCOMES:
1. Scale for Identification to the Symptom and Risks of Child Abuse and Neglect (SISRCAN) | Pretest
  This scale, consisting of 67 items in total, was developed to measure the knowledge levels of nurses and midwives about child abuse and neglect. This scale is a 5-point Likert type. The scale has 6 sub-dimensions. There are reverse scored items in the scale. The participant who answers all the items in the scale correctly is expected to get 335 full points. Each sub-dimension of the scale is evaluated by calculating the average score out of 5. The fact that the average score of the participants is close to 5 indicates that they answered the questions "correctly", and the closer to 1 indicates that they answered the questions "wrong". In the internal consistency analysis for reliability, the Cronbach alpha value was found to be 0.92.
1. Scale for Identification to the Symptom and Risks of Child Abuse and Neglect (SISRCAN) | Immediately after the intervention
  This scale, consisting of 67 items in total, was developed to measure the knowledge levels of nurses and midwives about child abuse and neglect. This scale is a 5-point Likert type. The scale has 6 sub-dimensions. There are reverse scored items in the scale. The participant who answers all the items in the scale correctly is expected to get 335 full points. Each sub-dimension of the scale is evaluated by calculating the average score out of 5. The fact that the average score of the participants is close to 5 indicates that they answered the questions "correctly", and the closer to 1 indicates that they answered the questions "wrong". In the internal consistency analysis for reliability, the Cronbach alpha value was found to be 0.92.
1. Scale for Identification to the Symptom and Risks of Child Abuse and Neglect (SISRCAN) | 1 month after the intervention
  This scale, consisting of 67 items in total, was developed to measure the knowledge levels of nurses and midwives about child abuse and neglect. This scale is a 5-point Likert type. The scale has 6 sub-dimensions. There are reverse scored items in the scale. The participant who answers all the items in the scale correctly is expected to get 335 full points. Each sub-dimension of the scale is evaluated by calculating the average score out of 5. The fact that the average score of the participants is close to 5 indicates that they answered the questions "correctly", and the closer to 1 indicates that they answered the questions "wrong". In the internal consistency analysis for reliability, the Cronbach alpha value was found to be 0.92.

CONTACTS AND LOCATIONS:
Overall Officials: Gokce Nz Cakir, BSN, Study Chair — Yeditepe University
Locations (1):
- Yeditepe University, Istanbul, Atasehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akcan, A., & Demiralay, Ş. (2016). Hemşirelik bölümü öğrencilerinin çocuk ihmal ve istismarına ilişkin algıları. Eğitim ve Öğretim Araştırmaları Dergisi, 5(32), 275-281.
- [Background] Altan, H. (2015). Üniversite Öğrencisi Gençlere Çocuk İstismarı Ve İhmali Konusunda Yapılan Eğitimin Bilgi Ve Farkındalıklarına Etkisi [Doktora, Gazi Üniversitesi].
- [Background] Austin AE, Lesak AM, Shanahan ME. Risk and protective factors for child maltreatment: A review. Curr Epidemiol Rep. 2020 Oct 7;7(4):334-342. doi: 10.1007/s40471-020-00252-3. PMID 34141519
- [Background] Bağ, Ö. F., & Bozkurt, G. (2021). Hemşirelerin Çocuk İhmal Ve İstismarina İlişkin Farkindaliklarini Etkileyen Faktörlerin İncelenmesi. Anadolu Hemşirelik Ve Sağlik Bilimleri Dergisi, 24(1), 17-24.
- [Background] Bahrami N, Tork-Torabi M, Sotoudeh R, Namnabati M. Perceived Child Abuse and Neglect in Hospitalized Children with Special Health Care Needs in Iran. Iran J Nurs Midwifery Res. 2021 Oct 22;26(6):526-530. doi: 10.4103/ijnmr.IJNMR_296_19. eCollection 2021 Nov-Dec. PMID 34900652
- [Background] Bakır, E., & Kapucu, S. (2017). Çocuk ihmali ve istismarının Türkiye'de yapılan araştırmalara yansıması: Bir literatür incelemesi. Hacettepe Üniversitesi Hemşirelik Fakültesi Dergisi, 4(2), 13-24.
- [Background] Başdaş, Ö., & Bozdağ, F. (2018). Hemşirelerin çocuk istismarı ve ihmalinin belirti ve risklerini tanılama durumlarının belirlenmesi. Mersin Üniversitesi Sağlık Bilimleri Dergisi, 11(3), 267-275.
- [Background] Burç, A., & Güdücü Tüfekci, F. (2015). Hemşirelerin çocuk istismarı ve ihmalinin belirti ve risklerini tanılama düzeyleri.
- [Background] Chen CJ, Chen YW, Chang HY, Feng JY. Screening Tools for Child Abuse Used by Healthcare Providers: A Systematic Review. J Nurs Res. 2022 Feb 1;30(1):e193. doi: 10.1097/JNR.0000000000000475. PMID 35050956
- [Background] Child Welfare Information Gateway. (2004). Risk and Protective Factors for Child Abuse and Neglect. U.S. Department of Health and Human Services, Administration for Children and Families, Children's Bureau. . https://www.childwelfare.gov/pubpdfs/riskprotectivefactors.pdf
- [Background] Child Welfare Information Gateway. (2019). What is child abuse and neglect? Recognizing the signs and symptoms. Washington, DC: U.S. Department of Health and Human Services, Children's Bureau.
- [Background] Cicchetti D. Socioemotional, Personality, and Biological Development: Illustrations from a Multilevel Developmental Psychopathology Perspective on Child Maltreatment. Annu Rev Psychol. 2016;67:187-211. doi: 10.1146/annurev-psych-122414-033259. PMID 26726964
- [Background] Conrad-Hiebner A, Byram E. The Temporal Impact of Economic Insecurity on Child Maltreatment: A Systematic Review. Trauma Violence Abuse. 2020 Jan;21(1):157-178. doi: 10.1177/1524838018756122. Epub 2018 Feb 4. PMID 29400135
- [Background] Erkut, Z., Gözen, D., & Beşirik, S. (2021). Hemşirelik Bölümü Son Sınıf Öğrencilerinin Çocuk İstismarı ve İhmalinin Belirti ve Risklerini Tanılamaya Yönelik Bilgi Düzeyleri ve Sosyodemografik Faktörlerle İlişkisi. Journal Education and Research in Nursing, 18(2), 231-240.
- [Background] Daley SF, Gonzalez D, Bethencourt Mirabal A, Afzal M. Child Abuse and Neglect. 2025 Apr 11. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK459146/ PMID 29083602
- [Background] Gubbels J, van der Put CE, Stams GJM, Assink M. Effective Components of School-Based Prevention Programs for Child Abuse: A Meta-Analytic Review. Clin Child Fam Psychol Rev. 2021 Sep;24(3):553-578. doi: 10.1007/s10567-021-00353-5. Epub 2021 Jun 4. PMID 34086183
- [Background] Jordan KS, Moore-Nadler M. Children at risk of maltreatment: identification and intervention in the emergency department. Adv Emerg Nurs J. 2014 Jan-Mar;36(1):97-106. doi: 10.1097/TME.0000000000000011. PMID 24487268
- [Background] Kuşlu, S., & Bulut, A. (2021). Çocuk İstismarı ve İhmaline Yönelik Hemşirelerin Bilgi, Tutum ve Davranışları: Literatür Taraması. Disiplinlerarası Çocuk Hakları Araştırmaları Dergisi, 1(2), 73-84.
- [Background] Külcü, D. P., & Karataş, H. (2016). Çocuk kliniklerinde çalişan hemşirelerin çocuk istismari ve ihmali konusunda bilgi düzeylerinin incelenmesi. Ege Üniversitesi Hemşirelik Fakültesi Dergisi, 32(1), 48-58.
- [Background] Ozbey, H., Ozcelep, G. A., Gul, U., & Kahriman, I. (2018). Knowledge and awareness of nursing students about child abuse and neglect. J Nurs Res Pract, 2(3), 21-25.
- [Background] Özçevik, D., Güneş, Ö. D., & OCAKÇI, A. F. (2018). Hemşirelik öğrencilerinin sosyo-kültürel ve demografik özelliklerinin çocuk istismarı ve ihmali farkındalığı ile ilişkisi. Ankara Sağlık Hizmetleri Dergisi, 17(2), 16-27.
- [Background] Poreddi V, Pashapu DR, Kathyayani BV, Gandhi S, El-Arousy W, Math SB. Nursing students' knowledge of child abuse and neglect in India. Br J Nurs. 2016 Mar 10-23;25(5):264-8. doi: 10.12968/bjon.2016.25.5.264. PMID 26972999
- [Background] Seferoğlu, E. G., Sezici, E., & Yiğit, D. (2019). Hemşirelik öğrencilerinin çocuk istismarı ve ihmalinin belirti ve risklerini tanılama düzeyleri. OPUS International Journal of Society Researches, 10(17), 257-276.
- [Background] Tek, S., & Karataş, G. (2021). Awareness Levels of Child Neglect and Abuse in Nursing Students. OPUS International Journal of Society Researches, 18(43), 6162-6176.
- [Background] Topçu, T. E., Erek Kazan, E., Küçük, S., Murat, Y., Alpaslan, B., Molozoğlu, H., & Özkan, B. (2022). Hemşirelik Öğrencilerinin Çocuk İstismarı ve İhmalinin Belirti ve Risklerini Tanılamaya İlişkin Bilgi Düzeyleri. Journal of Higher Education & Science/Yüksekögretim ve Bilim Dergisi, 12(2), 264-273.
- [Background] TUİK. (2021). Güvenlik Birimine Gelen veya Getirilen Çocuk İstatistikleri, 2020. Erişim adresi: https://data.tuik.gov.tr/Bulten/Index?p=Guvenlik-Birimine-Gelen-veya-Getirilen-Cocuk-Istatistikleri-2020-37200
- [Background] Yüksel, H., & Yüksel, M. (2014). Çocuk ihmali ve istismarı bağlamında Türkiye'de çocuk gelinler gerçeği. Çankırı Karatekin Üniversitesi Sosyal Bilimler Enstitüsü Dergisi, 5(2), 1-24.